CLINICAL TRIAL: NCT03523156
Title: Trachoma Elimination Study by Focused Antibiotic (TESFA): The Impact of an Enhanced Antibiotic Treatment Regimen on Trachoma in Amhara, Ethiopia
Brief Title: Trachoma Elimination Study by Focused Antibiotic (TESFA)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The Trachoma Elimination Study by Focused Antibiotic (TESFA): The Impact of an Enhanced Antibiotic Treatment Regimen on Trachoma in Amhara, Ethiopia is withdrawn due to severe delays and continued insecurity in the Amhara region of Ethiopia.
Sponsor: Emory University (Other)
Collaborators: The Carter Center (Other)
Responsible Party: Principal Investigator, Kelly Callahan, Program Director, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00085779
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Trachoma
Keywords: Antibiotics; Infectious diseases; Tropical medicine; Public health
MeSH Terms: conditions — Trachoma; Communicable Diseases | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Sixty-four kebeles (sub-districts) of Amhara will be randomized to receive annual mass treatment or annual mass treatment plus targeted treatment. One gott (village) per kebele will be selected and 50 children from each gott will be randomly selected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin mass treatment (Active Comparator): Persons living in regions randomized to this arm will receive mass drug administration (MDA) of azithromycin per the current annual MDA schedule.
  Interventions: Drug: Azithromycin mass treatment
- Azithromycin mass treatment plus targeted treatment (Experimental): In addition to azithromycin administration per the current annual MDA schedule, children in regions randomized to this arm will receive azithromycin targeted treatment.
  Interventions: Drug: Azithromycin mass treatment; Drug: Azithromycin targeted treatment

INTERVENTIONS:
Drug: Azithromycin mass treatment — Standard of care annual community-wide mass drug administration (MDA) will be provided at the normally scheduled time.
  Other Names: Zithromax
Drug: Azithromycin targeted treatment — Two rounds of treatment targeted to all children aged 2 to 9 years old. The first targeted round will be 1-2 weeks after the community-wide MDA and the second round will occur another 1-2 weeks later.
  Other Names: Zithromax
  Arms: Azithromycin mass treatment plus targeted treatment

SUMMARY:
The study population consists of all households residing in eligible kebeles (sub-districts) within districts in Amhara National Regional State which are identified as having a high prevalence of trachoma and infection measured from recent trachoma impact assessments. Within each study kebele, one village will be randomly selected to serve as the sentinel study site for that kebele. Once these villages are chosen, the study team will use government-provided census records, or perform a census in each village, and will randomly choose 50 children to serve as the sentinel children for the study. After the baseline visit, all kebeles will be randomized into one of the two treatment arms to either receive standard-or-care treatment, which is an annual community-wide mass drug administration (MDA), or the enhanced antibiotic treatment. Recruitment will take place at the selected children's household. Oral informed consent will be sought from village leader/chairmen before surveys are conducted in a village. Oral informed consent will then be obtained from household heads of those houses included in the study; and then from each participating individual. Oral consents will be obtained given the low literacy rates in rural Amhara.

Data collection will occur at baseline, week 4, month 12, and month 24 in both arms of the study. A head of household will be asked a series of household level questions, which will be followed by a household-level census, where all consenting participants residing in the selected households will have their eyes examined for trachoma signs. This is a non-invasive procedure whereby a trained trachoma grader flips each eyelid and examines for trachoma signs. Lastly, the selected child and one randomly selected adult will have their right eye lid swabbed for evidence of trachoma infection. The total estimated respondent burden is 30 to 45 minutes.

DETAILED DESCRIPTION:
Trachoma, caused by ocular infection with Chlamydia trachomatis, is one of the leading causes of preventable blindness worldwide with 51 countries known or suspected to be endemic for blinding trachoma. The World Health Organization (WHO) has recommended the Surgery, Antibiotic treatment, promotion of Facial cleanliness and hygiene, and Environmental improvement (SAFE) strategy for trachoma control. Annual mass drug administration (MDA) with the antibiotic azithromycin to treat trachoma is effective, at least in areas with moderate to low levels or trachoma. This has not been the experience in regions with high levels of trachoma including Amhara, Ethiopia. After 8 rounds of annual MDA, trachoma remains stubbornly high throughout the region. Given this experience from the Amhara region of Ethiopia, The Carter Center will work with local government partners at the regional, zonal, district, and sub-district levels to assess the effectiveness of a targeted antibiotic treatment regimen on trachoma prevalence by using a cluster randomized, controlled trial design with the understanding that increasing the need for drug in the short-term to intensify impact, may result in reduced need for drug in the long-term. The effectiveness of this alternative treatment regimen will be assessed over a period of 2 years by periodically evaluating trachoma outcomes throughout study communities.

The key objectives of this study are to:

1. To determine the effectiveness of an enhanced antibiotic treatment regimen characterized by a community-wide MDA followed by two rounds of targeted (to children age 2 to 9 years) treatment in quick succession (1-2 weeks apart) compared to annual standard-of-care MDA.
2. To determine the added cost and cost-effectiveness of an enhanced antibiotic treatment regimen compared to annual standard-of-care MDA.

ELIGIBILITY:
Cluster (kebele) Inclusion Criteria:

* The kebele must be located in Amhara and eligible for annual MDA with azithromycin under WHO treatment guidelines.
* Located within targeted districts where the prevalence of TF is high (at least 30%) and the prevalence of CT infection is suspected to be high (10% if possible) measured from the most recent trachoma impact assessment.
* The kebele representatives consent to participation in the trial.

Gott (village) Inclusion Criteria:

* At least 50 children residing in the gott.

Child Inclusion Criteria:

* Must reside in a cluster selected for this study.
* Must have a head of household or designated "adult-in-charge" who can provide consent for that child to be included in the study sample and to consent to allowing study staff to collect an ocular swab from the conjunctival epithelium.
* Child must assent to having a swab taken.
* Child must not have an ocular condition which would preclude grading trachoma or taking an ocular specimen.

Exclusion Criteria:

* none

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Chlamydia trachomatis (CT) infection | Month 12
  The community-level prevalence of CT infection in children aged 6 months to 9 years will be compared between study arms.

SECONDARY OUTCOMES:
Change in prevalence of trachomatous inflammation-follicular (TF) | Baseline, Week 4, Month 12, Month 24
  The prevalence of trachomatous inflammation-follicular (TF) among all household members will be noted at each visit and compared between study arms.
Change in prevalence of trachomatous inflammation-intense (TI) | Baseline, Week 4, Month 12, Month 24
  The prevalence of trachomatous inflammation-intense (TI) among all household members will be noted at each visit and compared between study arms.
Change in Chlamydia trachomatis (CT) infection in children | Baseline, Month 12, Month 24
  The change in prevalence of Chlamydia trachomatis (CT) infections in children ages 6 months to 9 years will be compared between study arms. Analysis will be conducted which will include all three of these time-points to compare infection prevalence between the comparison arms
Prevalence of Chlamydia trachomatis (CT) infection among adults | Month 12
  The prevalence of Chlamydia trachomatis (CT) infection among adults will be compared between study arms.
Cost | Month 24
  The cost of the enhanced intervention will be compared to the cost of the standard-of-care intervention.
Cost-effectiveness | Month 24
  The cost-effectiveness of the enhanced intervention will be compared to the cost of the standard-of-care intervention. The incremental cost effectiveness analysis ratio approach will be used. Effectiveness is defined as the percent CT reduction from baseline to 24 months and the outcome of this analysis will be the cost per percent of CT infection reduction.
Correlation between Chlamydial Infection and trachomatous inflammation-follicular (TF) and trachomatous inflammation-intense (TI) | Baseline, Week 4, Month 12, Month 24
  We will conduct cluster level analysis using cluster level Ct and clinical data including TF and TI.
Cluster-level Chlamydial load | Baseline, Week 4, Month 12, Month 24
  Infectious load for all individual specimens from children aged 6 months to 9 years who test positive for CT will be measured for chlamydia load. Chlamydial load will be noted at each visit and compared between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Callahan, MPH, Principal Investigator — The Carter Center